CLINICAL TRIAL: NCT06340386
Title: Italian Validation for the Female Sexual Function Index for Breast Cancer Patients (FSFI-BC)
Brief Title: Italian Validation of a Tool for Assessing Sexual Function After Breast Cancer, FSFI-BC
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1365
Record Dates: First submitted 2024-03-26; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with breast cancer and age <=50 years: Patients with diagnosis of breast cancer and age <=50 years
- Patients with breast cancer and age >50 years: Patients with diagnosis of breast cancer and age >50 years

SUMMARY:
This is a validation study of the italian language for the Female Sexual Function Index-Breast Cancer questionnaire.

The validation of the instrument in Italian will allow the identification of possible issues related to sexual health and enable the provision of adequate medical and psychosexual counseling to these patients, both in clinical practice and in research studies.

DETAILED DESCRIPTION:
The original version of the questionnaire will be validated in two phases: a) translation, b) reliability.

1. Translation of the items and administration to a small sample of volunteers to assess usability.

   In the first phase, the questionnaire will be translated following the 5 steps:
   1. forward translation by two independent translators (from English to Italian);
   2. synthesis (discussion between translators to resolve any discrepancies);
   3. backward translation (from Italian to English) by two additional independent translators;
   4. expert committee (translators, psychologists, sexology consultants) comparing the two versions of the questionnaire; 5) testing the first version of the questionnaire with a sample (N=20) of native Italian speakers to evaluate the adequacy of content and clarity of terms used and proceeding to the final version.
2. Reliability of the questionnaire. To assess the reliability of the questionnaire, it will be administered again after a 2-week interval to a smaller sample compared to the recruited patient sample.

ELIGIBILITY:
Inclusion Criteria:

1. Women with operable breast cancer;
2. Operated on between 2012 and 2020;
3. Randomly selected from the institutional database; 18 years of age (Age stratification: equally represented women aged <50 years and women aged ≥50 years);
4. Signing of the informed consent.

Exclusion Criteria:

1. Severe psychiatric or cognitive illness;
2. Ongoing psychological treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at European Institute of Oncology for a operable breast cancer between 2012 and 2020
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Validation of the italian translation of Female Sexual Function Index-Breast Cancer questionnaire | 12 months
  The measure of internal consistency utilized is Cronbach's alpha (α). The comparison will be done between the estimated α in the Italian questionnaire and the α of the original work.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy